CLINICAL TRIAL: NCT06525714
Title: Effect of Prophylactic Hyperthermic Intraperitonal Chemotherapy（HIPEC）After Radical Surgery on Long-term Survival for Locally Advanced Gastric Cancer（cT3N+M0 and cT4aN+/-M0）: A Randomized-controlled Study
Brief Title: Effect of HIPEC After Radical Surgery on Long-term Survival for Locally Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W100110120
Record Dates: First submitted 2024-07-25; First posted 2024-07-29 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer; Survival Rate
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomized-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cisplatin, oxaliplatin, tegafur. (Experimental): Cisplatin, oxaliplatin, tegafur.
  Interventions: Drug: cisplatin oxaliplatin tegafur

INTERVENTIONS:
Drug: cisplatin oxaliplatin tegafur — Within 48 hours postoperative, the first infusion was performed with 3000-4000 ml of saline and 50 mg/m2 cisplatin at 43°C, with an infusion rate of 600 ml/min for a duration of 2 hours. During treatment, close attention is given to the patient's heart rate, blood pressure, oxygenation, and other vital signs. A total of 2 HIPEC treatments were conducted, each 48 hours apart. Systemic chemotherapy is initiated 3-4 weeks postoperative for 6-8 cycles using SOX: intravenous injection of oxaliplatin (130 mg/m2) on the first day and oral administration of tegafur (40-60 mg twice daily, with doses adjusted for body surface area: <1.25 m2, 40 mg; 1.25m2 ≤ body surface area ≤ 1.5m2, 50mg; body surface area >1.5m2, 60 mg bid) from day 1 to 14.

SUMMARY:
The study focuses on patients with locally advanced gastric adenocarcinoma (cT3N+M0 and cT4aN+/-M0), assessing the feasibility, surgical safety, and oncological benefit of prophylactic HIPEC treatment following laparoscopic D2 radical surgery.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria will undergo laparoscopic D2 radical surgery. Before closing the abdomen during surgery, heat perfusion tubes are inserted, typically placing four tubes in a cross arrangement. Two drainage tubes at the pelvic floor exit through the upper abdomen, and two drainage tubes at the hepatorenal and splenorenal recesses exit through the lower abdomen, thus completing the tube placement.

Within 48 hours postoperative, the first infusion was performed with 3000-4000 ml of saline and 50 mg/m2 cisplatin at 43°C, with an infusion rate of 600 ml/min for a duration of 2 hours. During treatment, close attention is given to the patient's heart rate, blood pressure, oxygenation, and other vital signs. A total of 2 HIPEC treatments were conducted, each 48 hours apart. Systemic chemotherapy is initiated 3-4 weeks postoperative for 6-8 cycles using SOX: intravenous injection of oxaliplatin (130 mg/m2) on the first day and oral administration of tegafur (40-60 mg twice daily, with doses adjusted for body surface area: <1.25 m2, 40 mg; 1.25m2 ≤ body surface area ≤ 1.5m2, 50mg; body surface area >1.5m2, 60 mg bid) from day 1 to 14.

HIPEC is not performed postoperative. Systemic chemotherapy is initiated 3-4 weeks postoperative for 6-8 cycles using SOX: intravenous injection of oxaliplatin (130 mg/m2) on the first day and oral administration of tegafur (40-60 mg twice daily, with doses adjusted for body surface area: <1.25 m2, 40 mg; 1.25m2 ≤ body surface area ≤ 1.5m2, 50mg; body surface area >1.5m2, 60 mg bid) from day 1 to 14.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and ≤70 years;
2. Male or nonpregnant female;
3. Gastric adenocarcinoma cT3N+M0 and cT4aN+/-M0 (according to the 8th edition of the AJCC TNM staging system);
4. No distant metastasis, suitable for D2 lymph node dissection;
5. ECOG (Eastern Cooperative Oncology Group) performance status of 0-2;
6. No prior cytotoxic chemotherapy, radiotherapy, or immunotherapy;
7. Written informed consent given before any study-related procedures;

Exclusion Criteria:

1. Other cancers within the past 5 years;
2. Distant metastasis (M1) found during surgery;
3. ASA (American Society of Anesthesiologists) classification ≥IV and/or ECOG performance status >2;
4. Severe liver, kidney, cardiac, pulmonary, or coagulation dysfunction, or severe underlying diseases that make the patient unable to tolerate surgery;
5. A history of severe mental illness;
6. History of taking steroid medications;
7. Receiving other chemotherapy, radiotherapy, or immunotherapy;
8. Lack of written informed consent;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival rate | Three years after treatment
  Three-year overall survival after treatment

IPD SHARING:
Plan to Share IPD: No
There are plans to make individual participant data (IPD) available to other researchers. Includes only basic information such as name and gender.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Feng RM, Zong YN, Cao SM, Xu RH. Current cancer situation in China: good or bad news from the 2018 Global Cancer Statistics? Cancer Commun (Lond). 2019 Apr 29;39(1):22. doi: 10.1186/s40880-019-0368-6. PMID 31030667
- [Background] Saito H, Kono Y, Murakami Y, Kuroda H, Matsunaga T, Fukumoto Y, Tomohiro O, Fujiwara Y. Gross Appearance and Curability Are Predictive Factors of a Better Prognosis After Gastrectomy in Gastric Cancer Patients with Metastasis to the Adjacent Peritoneum of the Stomach. Yonago Acta Med. 2017 Sep 15;60(3):174-178. eCollection 2017 Sep. PMID 28959128
- [Background] Song H, Wang T, Tian L, Bai S, Chen L, Zuo Y, Xue Y. Macrophages on the Peritoneum are involved in Gastric Cancer Peritoneal Metastasis. J Cancer. 2019 Aug 29;10(22):5377-5387. doi: 10.7150/jca.31787. eCollection 2019. PMID 31632482
- [Background] Jo JC, Ryu MH, Koo DH, Ryoo BY, Kim HJ, Kim TW, Choi KD, Lee GH, Jung HY, Yook JH, Oh ST, Kim BS, Kim JH, Kang YK. Serum CA 19-9 as a prognostic factor in patients with metastatic gastric cancer. Asia Pac J Clin Oncol. 2013 Dec;9(4):324-30. doi: 10.1111/ajco.12019. Epub 2012 Nov 26. PMID 23176400
- [Background] Tustumi F, Bernardo WM, Dias AR, Ramos MF, Cecconello I, Zilberstein B, Ribeiro-Junior U. Detection value of free cancer cells in peritoneal washing in gastric cancer: a systematic review and meta-analysis. Clinics (Sao Paulo). 2016 Dec 1;71(12):733-745. doi: 10.6061/clinics/2016(12)10. PMID 28076519
- [Background] Sticca RP, Dach BW. Rationale for hyperthermia with intraoperative intraperitoneal chemotherapy agents. Surg Oncol Clin N Am. 2003 Jul;12(3):689-701. doi: 10.1016/s1055-3207(03)00029-2. PMID 14567025
- [Background] Rau B, Brandl A, Thuss-Patience P, Bergner F, Raue W, Arnold A, Horst D, Pratschke J, Biebl M. The efficacy of treatment options for patients with gastric cancer and peritoneal metastasis. Gastric Cancer. 2019 Nov;22(6):1226-1237. doi: 10.1007/s10120-019-00969-1. Epub 2019 May 7. PMID 31065877
- [Background] Yu HH, Yonemura Y, Ng HJ, Lee MC, Su BC, Hsieh MC. Benefit of Neoadjuvant Laparoscopic Hyperthermic Intraperitoneal Chemotherapy and Bidirectional Chemotherapy for Patients with Gastric Cancer with Peritoneal Carcinomatosis Considering Cytoreductive Surgery. Cancers (Basel). 2023 Jun 29;15(13):3401. doi: 10.3390/cancers15133401. PMID 37444511
- [Background] Hung HC, Hsu PJ, Lee CW, Hsu JT, Wu TJ. Cytoreductive Surgery with Hyperthermic Intraperitoneal Chemotherapy for Gastric Cancer with Peritoneal Carcinomatosis: Additional Information Helps to Optimize Patient Selection before Surgery. Cancers (Basel). 2023 Mar 31;15(7):2089. doi: 10.3390/cancers15072089. PMID 37046754
- [Background] Zhong Y, Kang W, Hu H, Li W, Zhang J, Tian Y. Lobaplatin-based prophylactic hyperthermic intraperitoneal chemotherapy for T4 gastric cancer patients: A retrospective clinical study. Front Oncol. 2023 Jan 18;13:995618. doi: 10.3389/fonc.2023.995618. eCollection 2023. PMID 36741012
- [Background] Zhang J, Sun Y, Bai X, Wang P, Tian L, Tian Y, Zhong Y. Single versus multiple hyperthermic intraperitoneal chemotherapy applications for T4 gastric cancer patients: Efficacy and safety profiles. Front Oncol. 2023 Mar 17;13:1109633. doi: 10.3389/fonc.2023.1109633. eCollection 2023. PMID 37007142
- [Background] Bazarbashi S, Badran A, Gad AM, Aljubran A, Alzahrani A, Alshibani A, Alrakaf R, Elhassan T, Alsuhaibani A, Elshenawy MA. Combined Prophylactic Hyperthermic Intraperitoneal Chemotherapy and Intraoperative Radiotherapy for Localized Gastroesophageal Junction and Gastric Cancer: A Comparative Nonrandomized Study. Ann Surg Oncol. 2023 Jan;30(1):426-432. doi: 10.1245/s10434-022-12467-3. Epub 2022 Aug 30. PMID 36042103